CLINICAL TRIAL: NCT05843591
Title: Effects of Aerobic Exercise or Tai Chi Chuan Interventions on Problematic Mobile Phone Use and the Potential Role of Intestinal Flora: a Multi-arm Randomized Controlled Trial
Brief Title: Exercise Interventions on Problematic Mobile Phone Use: a Multi-arm Randomized Controlled Trial
Status: Completed | Type: Observational
Sponsor: Anhui Medical University (Other)
Responsible Party: Principal Investigator, Kexin Zhang, professor, Anhui Medical University
Other Study IDs: KZhang
Record Dates: First submitted 2023-04-25; First posted 2023-05-06 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-04

CONDITIONS: Exercise Intervention; Tai Chi Chuan; Intestinal Flora; Randomized Clinical Trial
Keywords: Problematic Mobile Phone Use; Exercise Intervention; Aerobic Exercise; Tai Chi Chuan; intestinal flora
MeSH Terms: interventions — Exercise; Tai Ji

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Aerobic Exercise group: Participants in the aerobic exercise (AE) group were asked to perform moderate to high intensity regular aerobic exercise. Exercise was required 3 times per week for at least 1 hour each time. At the beginning of the exercise, they were required to sign in at the research personnel, and at the end of the exercise, they were also required to sign out at the research personnel. However, there was no restriction on the type of exercise, which could be running, basketball, badminton, table tennis, tennis, rope skipping, dancing, etc.; there was no restriction on the form of exercise, which could be individual or group exercise; there was no restriction on the period of exercise start, which could be any time of the day to start exercise.
  Interventions: Behavioral: aerobic exercise or Tai Chi Chuan interventions
- Tai Chi Chuan group: Participants in the Tai Chi Chuan (TCC) group attended an 8-week Tai Chi training program, which consists of 24-form Tai Chi and Bafa Wubu of Tai Chi. Certified instructors administer and guide Tai Chi Chuan activities. We set up 6 Tai Chi Chuan classes each week, and participants in the Tai Chi Chuan group can participate in any 3 of the 6 classes each week to be considered as completing the task. Each 1-hour training session consists of a brief warm-up stretching session followed by standard Tai Chi routine activities.
  Interventions: Behavioral: aerobic exercise or Tai Chi Chuan interventions
- Wait-List Control group: Participants in the wait-list control (WLC) group received no intervention in addition to their usual physical education classes.
  Interventions: Behavioral: aerobic exercise or Tai Chi Chuan interventions

INTERVENTIONS:
Behavioral: aerobic exercise or Tai Chi Chuan interventions — 8-week aerobic exercise (AE group), 8-week Tai Chi Chuan training (TCC group)
  Other Names: aerobic exercise; Tai Chi Chuan

SUMMARY:
Problematic mobile phone use (PMPU) has been described as a growing public health issue. This randomized controlled trial aimed to determine if aerobic exercise or Tai Chi Chuan as compared to the wait-list control group decreased PMPU-related symptoms; and to analyze the composition of the intestinal flora in the three study groups to explore the correlation between PMPU scores and flora species. A consecutive sample of 90 college students with PMPU was randomized to the aerobic exercise group (AE group, n = 30), the Tai Chi Chuan group (TCC group, n = 30), or the wait-list control group (WLC group, n = 30). The primary outcome was addiction symptoms, i.e., the PMPU score as assessed by the Smartphone Addiction Scale-Short Version (SAS-SV). Secondary outcomes were the emotion-related symptoms (depression, anxiety, self-esteem and self-efficacy), and physical-related symptoms (sleep quality, physical-fatigue and mental-fatigue). Intervention effects were analyzed via generalized estimated equation analysis (GEE).

ELIGIBILITY:
Inclusion Criteria:

* (1) be 18 years or older; (2) college students; (3) fulfill the Smartphone Addiction Scale-Short Version (SAS-SV) criteria for PMPU; (4) have a low level of daily physical activity.

Exclusion Criteria:

* (1) regular practice of moderate and higher intensity exercise (Physical activity was measured using the Physical Activity Rating Scale-3 (PARS-3), which is a 3-item self-reported scale comprising intensity, duration and frequency [14]. Exercise was considered to be of more than moderate intensity when the PARS-3 scores was >42); (2) any major disease (cardiovascular disease, respiratory illness, and musculoskeletal disorder) that can affect them to participate in exercise training; (3) any gastrointestinal diseases and other diseases affecting intestinal bacteria; and (4) any severe mental illness (e.g., depression, anxiety, bipolar disorder, obsessive-compulsive disorder, eating disorder, and post-traumatic stress disorder).

Ages: 18 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Participants were recruited between February 2022 and March 2022. Participants from Anhui Medical University were recruited through promotion in academic departments and student societies as well as advertisements in social media (We-chat and QQ). The coordinator subsequently contacted potential participants via We-chat to provide them with information regarding the study; and determine their interest and eligibility.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2022-02-04 (Actual); Primary Completion 2022-06-03 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Smartphone Addiction Scale-Short Version (SAS-SV) | 2 months
  Problematic mobile phone use levels

SECONDARY OUTCOMES:
Zung's Self Rating Depression Scale (SDS) | 2 months
  Depression levels
Zung's Self-Rating Anxiety Scale (SAS) | 2 months
  Anxiety levels
Rosenberg self-esteem scale (RSES) | 2 months
  Self-esteem levels
General Self-Efficacy Scale (GSES) | 2 months
  Self-Efficacy levels
Pittsburgh Sleep Quality Index (PSQI) | 2 months
  Sleep Quality levels
Fatigue Scale-14 | 2 months
  physical and mental fatigue levels
Intestinal flora | 2 months
  Fecal microbial DNA was extracted using the QIAamp Fast DNA Stool Mini kit (Qiagen, Hilden, Germany) according to the manufacturer's instructions. All procedures of DNA extraction were performed in a class II biosafety cabinet. Universal primers (341F and 805R) linked with indices and sequencing adaptors were used to amplify the V3-V4 regions of the 16S rRNA gene. The amplification products were detected by agarose gel electrophoresis, and the amplification products were purified by nucleic acid purification beads to obtain the original library of the sample. The library quality was assessed on the Agilent Bioanalyzer 2100 system. The 16S rRNA gene amplification products sequencing was performed with the 2 × 250 bp paired-end method using the Illumina MiSeq Benchtop Sequencer [48] at the Genesky Biotechnologies Inc. (Shanghai, China).

CONTACTS AND LOCATIONS:
Locations (1):
- Anhui Medical University, Hefei, Anhui, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhang K, Guo H, Zhang X, Yang H, Yuan G, Zhu Z, Lu X, Zhang J, Du J, Shi H, Jin G, Ren J, Hao J, Sun Y, Su P, Zhang Z. Effects of aerobic exercise or Tai Chi Chuan interventions on problematic mobile phone use and the potential role of intestinal flora: A multi-arm randomized controlled trial. J Psychiatr Res. 2024 Feb;170:394-407. doi: 10.1016/j.jpsychires.2024.01.012. Epub 2024 Jan 8. PMID 38218013